CLINICAL TRIAL: NCT03776890
Title: DeStress for Health: Partnering With Granville and Vance Counties to Reduce Stress and Cancer Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00100183
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2020-03

CONDITIONS: Stress Reduction
Keywords: stress reduction; rural; health behaviors; north carolina
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DeStress for Health Program Participants (Experimental): Rural residents 18 years and older of Granville and Vance counties (n=30) will be recruited to participate.
  Interventions: Behavioral: DeStress for Health Program

INTERVENTIONS:
Behavioral: DeStress for Health Program — The program will consist of 4 in person sessions that are based on empirically supported Positive Psychosocial Well-Being PPWB components including Optimism, Mindfulness, Positive Reprisal as well as Strengths-based Cognitive Behavioral Therapy (SBCBT) to improve behavioral self-regulation towards health-related goals. Research staff will conduct face-to-face surveys with participants at baseline and at end of program. Finally, we will conduct a phone-based survey 30 days after program completion to assess sustainability of intervention effects.

SUMMARY:
The purpose of this research study is to determine whether a positive psychology intervention paired with a health behavior intervention is successful in decreasing perceived stress and increasing positive affect in residents of Vance and Granville County. Participants will attend 4 classes that occur once a week. The first class will focus on nutrition, the second class will focus on exercise, the 3rd class will focus on tobacco use, and the 4th class that will review the previous 3 classes and help participants incorporate the strategies taught in the Destress for Health Program into their everyday lives. The duration of each class is 1 hour and the classes will be held once a week for a total of 4 weeks. Participants in this research study will be asked to complete 2 surveys. The first survey will occur during class 1, and will ask participants about their demographic information, health behaviors, stress levels, emotions, and behaviors. The second survey will be conducted over the phone and will occur 30-days after the final class and will ask participants about their health behaviors, stress levels, emotions, behaviors and also about whether or not they felt the classes they attended were useful to them. Total study duration is about 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Live in Granville or Vance Counties;
* >18 years old;
* Interested in participating a stress reduction study
* Speak English

Exclusion Criteria:

* Does Not Live in Granville or Vance Counties
* Under 18 years of age
* Not interested in participating in a stress reduction study
* Does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants Recruited in a 6-Month Time-frame | 6 Months
  Measured via subject enrollment log
Percentage of Participants That Stay in Study for Duration | 3 Months
  Measured via subject enrollment log
Percentage of Participants That Attend All Intervention Sessions | 3 Months
  Measured via subject enrollment log
Percent of Participants Rating Intervention as Useful | 3 Months
  Measured on a scale from 1-5 with 1 being "Not Useful at All" and 5 being "Extremely Useful".
Percent of Participants Recommending Intervention to Friend | 3 Months
  Measured on a scale from 1-5 with 1 being "Not at All" and 5 being "Extremely".

SECONDARY OUTCOMES:
Change in Stress Self Regulation As Measured By a Survey | Baseline, 3 Months
Change in Positive Emotion As Measured by a Survey | Baseline, 3 Months
Change in Behavioral Self Regulation As Measured by a Survey | Baseline, 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Devon Noonan, Ph.D, Principal Investigator — Duke School of Nursing
Locations (1):
- Granville Vance Public Health Department, Oxford, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No